CLINICAL TRIAL: NCT02148354
Title: Differential Efficacy of an Internet Delivered Intervention Program for the Prevention and Treatment of Mild to Moderate Depression With or Without Support by the Therapist
Brief Title: Internet Delivered Intervention Program for the Prevention and Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2014-03-13; First posted 2014-05-28 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Internet-based Treatment for Depression
Keywords: Depression; Self-applied treatment; Internet; Support by the therapist; Cognitive-Behavioural Treatment; Positive Psychology; Behavioral Activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group with support by the therapist. (Experimental): Intervention group that do the Smiling is Fun program and receives support by the therapist (a brief weekly two-minute call without clinical content).
  Interventions: Behavioral: Smiling is Fun
- Group without support by the therapist (Experimental): Intervention group that do the Smiling is Fun program and does not receive support by the therapist.
  Interventions: Behavioral: Smiling is Fun
- Waiting list control group (Other): Control group that could access the Smiling is Fun program after waiting for 12 weeks.
  After that time, those participants still interested were randomly assigned to one of two intervention conditions (with or without support by the therapist).
  Interventions: Behavioral: Smiling is Fun

INTERVENTIONS:
Behavioral: Smiling is Fun — Smiling is Fun is an internet-delivered self-help program for emotional disorders, which will allow the individual to learn and practice adaptive ways to cope with depression and daily problems. The program includes eight modules: Motivation for change, Understanding emotional problems; Learning to move on; Learning to enjoy; Learning to live; Living and learning and From now on, what else…?. Furthermore the program uses three transversal tools: 1) Activity report for self-monitoring, whose aim is to provide feedback to the user and help him see that his mood is related to the activities performed, 2) The calendar, and 3) "How am I?" offers a set of graphs and feedbacks to chart the user's progress.
  Other Names: Coping withs stress; Emotion Regulation Program

SUMMARY:
The purpose of this study is to determine the differential effectiveness of a self applied treatment delivered via Internet for the prevention and treatment of depression, with or without support by the therapist, compared to a waiting list control group. The principal hypothesis is that the two intervention groups will improve significantly compared to the waiting list control group, and without significant differences between them. The investigators believe that the support of ICTs may be doing a similar function as the weekly support call (to offer feedback, to reinforce, to motivate the participants, etc.). Furthermore the investigators hypothesize that the intervention program will be a useful tool for a secondary and tertiary prevention of depression.

DETAILED DESCRIPTION:
It is know that 25% of all human beings will suffer from depression at any moment over their lives and it will become one of the three leading causes of disability in 2030 (Mathers and Loncar, 2006). A very important challenge today consists on addressing the issue of depression from a preventive perspective (Mihalopoulos and Vos, 2013) operating in each of its three levels: primary prevention, to reduce its incidence, secondary prevention, for people who have some risk factor or those who show subclinical symptoms, and tertiary prevention, to minimize the limitations caused by an already established disorder (Commission on Chronic Illness, 1957; Vazquez and Torres, 2007). As Cuijpers, Beekman et al. (2012) point out in a recent paper, it is important to develop better strategies and tools to identify individuals at risk and the design of prevention programs. The investigators have evidence based psychological treatments for depression (Nathan and Gorman, 2007) and, although less there are also interventions focusing on its prevention (Cuijpers et al., 2008, Horowitz y Garber, 2006; Muñoz et al., 2010). However, they have an important limitation: the provision of mental health services is generally less than adequate in terms of accessibility and quality (Hinrichsen, 2010, Institute of Medicine, 2008; Kazdin and Blase, 2011). The Information and Communication Technologies (ICTs), especially the use of the Internet to support the implementation of the interventions (treatment or prevention), have proven to be a powerful means for its effective deployment in general mental healthcare provision. Although data using Internet-based interventions are consistent and promising, there are still important problems to solve: not all patients continue and complete these programs. The meta-analysis of studies on Internet-based treatments for depression report a dropout rate of 32% (range 0-75%) (Kaltenthaler, Parry, Beverley and Ferriter, 2008; Melville, Casey and Kavanagh, 2010). This problem could have various causes and one of which may be the fact of providing or not human support (Andersson et al., 2009). Recently, there has been increased research to determine the importance of human support in such interventions (Richards y Richardsson, 2012; Hilvert-Bruce, Rossouw, Wong, Sunderland and Andrews, 2012). The studies of meta-analysis find that the Internet-based treatments, in which support is given throughout the implementation of the program, produce greater effect sizes and less dropout rates than Internet-based programs without any human support (Andersson and Cuijpers, 2009; Richards and Richardson, 2012). It is important to note that the majority of studies mean support when it is administered by a person (therapist, consultant or researcher) and not by the ICTs (automated reminders, e-mails or mobile SMS) (Richards and Richardson, 2012). Now, there has also been recent evidence of the effectiveness of the self-applied treatments without any contact or support from a therapist, consultant or researcher (Cuijpers, Donker et al, 2011). Nevertheless, there are still few randomized controlled trials that specifically examine this issue (Berger et al., 2011, Clarke et al, 2005; Farrer, Christensen, Griffiths and Mackinnon, 2011). This is the principal objective of the present work, given the importance that this may have for the future developments in this field. The investigators addressed: It is necessary a weekly support call from a therapist during the course of an Internet- based intervention program, or is it enough just the support of the ICTs?. Because of this, the investigators have developed an Internet-based program (Smiling is Fun) for the prevention and treatment of depression (mild to moderate), and have carried out a randomized controlled trial with three experimental conditions: a) Intervention group with human support (two minutes weekly support call without clinical content); b) Intervention group without human support; c) Waiting list control condition. The two intervention groups received automated support from the ICTs: two weekly automated mobile phone messages, reminding of the importance of doing the tasks proposed by the program and, an automated e-mail encouraging them to continue with the modules in case they have not accesses the program for a week. The principal hypothesis is that the two intervention groups will improve significantly compared to the waiting list control group, and without significant differences among themselves. The investigators believe that the support of ICTs may be doing a similar function as the weekly support call (to offer feedback, to reinforce, to motivate the participants, etc.). Furthermore the investigators hypothesize that the intervention program will be a useful tool for a secondary and tertiary prevention of depression.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* Be willing to participate in the study.
* Be able to use a computer and having an Internet connection at home.
* Be able to understand and read Spanish.
* Minimal, mild, or moderate depression (score no more than 28 in the BDI-II).
* Experience, at least, one stressful event in their lives that provokes them an interference.

Exclusion Criteria:

* Be receiving psychological treatment.
* Have received another psychological treatment in the past year.
* A severe mental disorder on Axis I: abuse or dependence of alcohol or other substances, psychotic disorder or dementia.
* Presence of suicidal ideation or plan (Evaluated by MINI and item 9 of the BDI-II).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from Beck Depression Inventory II (BDI-II) at 3, 6 and 12 months follow-ups | Up to 12 months
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and test-retest reliability of around 0.8. The Spanish version of this instrument has also shown a high internal consistency (Cronbach's alpha of 0.87) for both the general and the clinical population (Cronbach's alpha of 0.89). Summed to obtain the total score, which can be a maximum of 63 points. According to the BDI-II manual scores of 0 to 13 denote minimal depression, scores of 14 to 19 denote mild depression, scores of 20 to 28 denote moderate depression and over 28 indicates severe depression.

SECONDARY OUTCOMES:
Change from Positive and Negative Affect Scale (PANAS) at 3, 6 and 12 months follow-ups | Up to 12 months
  PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is 10 to 50. The Spanish version has demonstrated high internal consistency (0.89 to 0.91 for PA and NA in women and 0.87 for AP and 0.89 for AN in men) in college students. This is consistent with the findings in the literature.
Change from Overall Anxiety Severity and Impairment Scale (OASIS) at 3, 6 and 12 months follow-ups | Up to 12 months
  OASIS consists of 5 items that measure the frequency and severity of anxiety, as well as the level of avoidance, work/ school/home interference, and social interference associated to anxiety. A psychometric analysis of the OASIS scale found good internal consistency (Cronbach's alpha = 0.80), test-retest reliability (k = 5.82) and convergent validity for this scale.
Change from Overall Depression Severity and Impairment Scale (ODSIS) at 3, 6 and 12 months follow-ups | Up to 12 months
  ODSIS is a self-report measure which consists of 5 items, evaluating experiences related to depression. ODSIS measures the frequency and severity of depression, as well as the level of avoidance, work/school/home interference, and social interference associated to depression. So far, no other studies examining the psychometric properties of this scale have been published. It is recommended to use and to interpret it in the same way that OASIS.

OTHER OUTCOMES:
Change from Multicultural Quality of Life Index (MQLI) at 3, 6 and 12 months follow-ups | Up to 12 months
  It is a self-administered questionnaire that uses 10 items to assess global perception of quality of life in addition to physical and emotional well-being, self-care, occupational, and interpersonal functioning, community and services support, and personal and spiritual fulfilment. The homogeneity of the questionnaire proved to be good, yielding a Cronbach's alpha coefficient of 0.79 and has applicability, reliability, and validity.
Change from Perceived Stress Scale (PSS) at 3, 6 and 12 months follow-ups | Up to 12 months
  The PSS is a 14-item self-report questionnaire that assesses the degree to which recent life situations are appraised as stressful. Spanish validation of this scale has an internal consistency of 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, Professor, Study Director — University Jaume I, Castellón, Spain
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Botella C, Mira A, Garcia-Palacios A, Quero S, Navarro MV, Riera Lopez Del Amo A, Molinari G, Castilla D, Moragrega I, Soler C, Alcaniz M, Banos RM. Smiling is fun: a Coping with Stress and Emotion Regulation Program. Stud Health Technol Inform. 2012;181:123-7. PMID 22954841
- [Background] Mira A, Botella C, García-Palacios A., Riera A, Quero S, Alcañiz M, Baños RM. An Internet-based Program to Cope with Regulating Stress and Emotion: An Example of Positive Technology. Journal of Cybertherapy & Rehabilitation, 2(1): 22-23, 2012.
- [Background] Mira A, Botella C, García-Palacios A, Bretón-López J, Moragrega I, Riera-López del Amo A, Quero S, Pérez-Ara, MA, Baños RM. Coping with Stress: A Program for the Prevention of Depression. Information and Communication Technologies applied to Mental Health. Proceedings of the 1st Workshop on ICT applied to Mental Health, 48-52, 2012
- [Background] Alcañiz, M, Zaragoza I, Rey B, Botella C, Moragrega I, Baños RM. Personal Health Systems: The OPTIMI Project. Journal of Cybertherapy & Rehabilitation 1: 20-23, 2011.
- [Derived] Mira A, Breton-Lopez J, Enrique A, Castilla D, Garcia-Palacios A, Banos R, Botella C. Exploring the Incorporation of a Positive Psychology Component in a Cognitive Behavioral Internet-Based Program for Depressive Symptoms. Results Throughout the Intervention Process. Front Psychol. 2018 Nov 29;9:2360. doi: 10.3389/fpsyg.2018.02360. eCollection 2018. PMID 30555384
- See also: Laboratory of Psychology and Technology of the University Juame I — http://www.labpsitec.uji.es
- See also: American Psychological Association — http://www.apa.org
- See also: National Institute for Health and Clinical Excellence — http://www.nice.org.uk